CLINICAL TRIAL: NCT01166490
Title: A Phase 1, Open-Label, Dose Escalation Study of ASG-5ME in Patients With Pancreatic or Gastric Adenocarcinoma
Brief Title: A Phase 1 Dose Escalation Trial of ASG-5ME in Pancreatic or Gastric Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASG5ME-002
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Gastric Neoplasms; Pancreatic Neoplasms
Keywords: Monomethyl auristatin E (MMAE); Immunotherapy; AGS-5 Antigen; SLC44A4 Antigen; Gastric Neoplasms; Pancreatic Neoplasms; Antibody-Drug Conjugate; Antibodies, Monoclonal; Drug Therapy
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — ASG-5ME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ASG-5ME
  Interventions: Drug: ASG-5ME

INTERVENTIONS:
Drug: ASG-5ME — 0.3-3.0 mg/kg IV on Days 1, 8, and 15 of 28-day cycles

SUMMARY:
This is a phase 1, open-label, dose-escalation clinical trial to evaluate the safety and tolerability of ASG-5ME and identify the maximum tolerated dose in patients with pathologically confirmed metastatic pancreatic adenocarcinoma, and to evaluate safety and tolerability in patients with relapsed or refractory gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic pancreatic adenocarcinoma or pathologically confirmed AGS-5-positive gastric or gastric esophageal junction adenocarcinoma
* Measurable disease (at least one nonresectable, non-nodal lesion greater than or equal to 10 mm in longest diameter or nodal lesion greater than or equal to 15 mm in shortest axis)
* ECOG performance status of 0 or 1
* May be untreated or have previously received treatment for pancreatic adenocarcinoma or must have relapsed or refractory disease following 1 prior systemic therapy for metastatic gastric adenocarcinoma. For patients who have previously received treatment, it must be at least 2 weeks since the last systemic therapy or radiation, and at least 4 weeks since treatment with any monoclonal antibody (other than bevacizumab).

Exclusion Criteria:

* Evidence or history of central nervous system metastases
* History of another primary malignancy that has not been in remission for at least 3 years
* Documented history of a cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms consistent with NYHA Class III-IV within 6 months prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | Through 1 month after last dose

SECONDARY OUTCOMES:
Best clinical response | Every 2 months
Overall and progression-free survival | Every month until death or study closure
Concentrations of ASG-5ME and metabolites in blood | Through 1 month after last dose
Incidence of antitherapeutic antibodies in blood | Through 1 month after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, BCOP, Study Director — Seagen Inc.
Locations (7):
- United States (7):
  - TGen Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - University of California at San Francisco, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington